CLINICAL TRIAL: NCT07011082
Title: Hair Biomarkers Study
Acronym: HBS-II
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kanwaljeet Anand, Director of Stanford Child Wellness Lab, Stanford University
Other Study IDs: IRB-71555; 2R01HD099296-05 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Toxic stress; Infants; Cortisol; Oxytocin; Early child development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Infants: Ages between 6-24 months
  Interventions: Other: Stress preventative measures
- Healthy Mothers: Mothers with children aged between 6-24 months who are eligible for the HBS-II
  Interventions: Other: Stress preventative measures

INTERVENTIONS:
Other: Stress preventative measures — These studies will address fundamental gaps in our current knowledge and establish a scientific framework to investigate the long-term effects of early childhood adversity, physical or emotional trauma, child maltreatment, or other adverse experiences in early childhood, as well as the preventive and protective effects of loving, nurturing, and consistent caregiving offered to young children during their early childhood

SUMMARY:
Young children aged 0-4 years may be exposed to adverse childhood experiences (ACEs) and/or early life adversity (ELA), which are linked with worse physical and mental health across their lifespan. On the other hand, positive childhood experiences (PCEs) can build resilience and prevent or protect against these detrimental outcomes. Data analyses will assess the interactions of ACEs, PCEs, parenting, and poverty on the early social psychology of childhood and develop objective measures for altered stress regulation using hair cortisol as a chronic stress biomarker.

DETAILED DESCRIPTION:
To elucidate the longitudinal changes underlying HPA-axis dysregulation, using community-based participatory research (CBPR) methods, the investigators have designed a prospective longitudinal study to enroll children aged 6-24 months from families living within Santa Clara, San Mateo, and Alameda Counties. This study will enroll 600 healthy children (as defined by the American Academy of Pediatrics) and each child will be assessed 5 times at 6-month intervals for a total of 2 years.

The investigators will collect serial hair samples at each visit, obtain anthropometric measures at yearly intervals, and also assess the child's cognitive, behavioral, social-emotional, relational, and other outcomes using bilingual parental surveys.

Parents will also provide basic demographic data, other parent- and family-related factors via bilingual questionnaires. Parents have the option of refusing to answer any question or complete the survey instruments that they are not comfortable with completing. The questionnaires that will be used in this study are the Demographics and Child Relationships Survey, the Child Opportunity Index 2.0 (SDOH), the Parenting Stress Scale (PSS), the Brief Symptom Inventory (BSI-18), the Conner-Davidson Resilience Index (CD-RISC-10), the Interfaith Spirituality Scale - Short Form (IFS-SF), the Health Mindset Questionnaire, and Parenting Styles & Dimensions Questionnaire for parents; as well as the Child Health History Survey (CHHx), the Ages and Stages Questionnaire (ASQ-3), the ASQ Social Emotional Questionnaire (ASQ:SE-2), the Speech & Language Assessment Scale (SLAS), the Child Aces & Related Life Events Scale (PEARLS 2.0), the BRIEF-Preschool Executive Functions Scale, the Positive Childhood Experiences Scale (PCEs), and the Child Flourishing Index for their child. At Study Exit, the parents will be asked to complete a very brief Study Closeout Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy children aged 6 months to 24 months and their mothers (or father, if mother is not able to participate).
2. Living in Santa Clara County, San Mateo County, or Alameda County in Northern California.
3. Willing to give their home address (in order to receive the study kits at home).
4. Committed to regular follow-up at 6-month intervals for the full study duration of 2 years.

Exclusion Criteria:

1. Children with tinea capitis, alopecia areata, scalp eczema, dermatitis, or other scalp conditions.
2. Children exposed to systemic steroid therapy for any diagnosis in the 3 months prior to study entry.
3. Children receiving any other prescription drugs that alter HPA axis function or cortisol release, if the period of exposure is 2 weeks or longer within the 3 months prior to study entry.
4. Children with chronic medical conditions such as cystic fibrosis, sickle cell disease, asthma, eczema, or other chronic conditions.
5. Children with known developmental delay, Trisomy-21 and other chromosomal anomalies, seizure disorders, chronic pain, cerebral palsy, or other disabilities.
6. Children whose hair has received chemical exposures (e.g., dying, bleaching, chemical straightening, perming) in the 90 days prior to study entry or for 90 days before each follow-up appointment during the 2-year study period.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Normal, healthy children aged 6 months to 24 months and their biological mothers (or father, if mother is not able to participate), in order to study the impact of early social ecology on their nascent social psychology, growth, and development in early childhood.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Identification of Participants hair cortisol concentrations (HCC) and hair oxytocin concentrations (HOC) | Hair samples measured at study entry and 6 month intervals up to 2 years (Study entry, 6-month, 12-month, 18-month, 24-month)
Hair Cortisol Concentration (HCC), nanograms cortisol/milligram of hair | From enrollment to end of study in 2 years
Hair Oxytocin Concentration (HOC), picogram oxytocin/milligram of hair | From enrollment to end of study in 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of proprietary methods used for analysis of hair samples.